CLINICAL TRIAL: NCT06921434
Title: Comparative Evaluation of Monk Fruit and Splenda on Salivary ph and Streptococcus Mutans Growth (an in Vivo Study)
Brief Title: the Effect of Monk Fruit and Splenda on Salivary Ph and Streptococcus Mutans Count in Vivo Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Kawthar Salman Alharan, master student, Al-Mustansiriyah University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mustansiriyah U
Record Dates: First submitted 2025-04-01; First posted 2025-04-10 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Caries Active
MeSH Terms: interventions — trichlorosucrose

STUDY DESIGN:
Intervention Model Description: parallel Assignment 90 participants will divided into 3 groups (Monk fruit ,Splenda ,and control group sucrose)and each group will receive only one intervention without switching
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- monk fruit sweetener group 30 participants (Experimental)
  Interventions: Dietary Supplement: Monk fruit sweetener mouth rinse
- Splenda (sucralose) sweetener group 30 participants (Experimental)
  Interventions: Dietary Supplement: Splenda (sucralose) sweetener mouth rinse
- positive control group (sucrose) 30 participants (Active Comparator)
  Interventions: Dietary Supplement: Sucrose mouth rinse

INTERVENTIONS:
Dietary Supplement: Monk fruit sweetener mouth rinse — monk fruit mouth rinse 10 grams of sweetener powder and 90 ml of distilled water for 30 participants for 1 minute
  Arms: monk fruit sweetener group 30 participants
Dietary Supplement: Splenda (sucralose) sweetener mouth rinse — 10 g of splenda powder with 90 ml of distilled water for 30 participants for 1 minute
  Arms: Splenda (sucralose) sweetener group 30 participants
Dietary Supplement: Sucrose mouth rinse — 10 g of sucrose powder dissolved in 90 ml of distilled water as a positive control group for 30 participants for 1 minute
  Arms: positive control group (sucrose) 30 participants

SUMMARY:
This study aims to evaluate the changes in salivary pH and Streptococcus mutans count by preparing a solution containing these sweeteners dissolved in distilled water and administering it to the participants. Saliva samples will be collected before using the mouth rinse, and salivary pH will be measured using a pH meter, while S. mutans count will be analyzed in the laboratory.

After consuming the solution, salivary pH will be assessed at 1 minute, 15 minutes, and 30 minutes, while the growth of S. mutans will be examined 30 minutes post-rinse.

DETAILED DESCRIPTION:
90 participants who meet the inclusion criteria-having no active caries, aged between 20 and 24 years, and not taking medications that affect saliva-will be included in the study. They will be divided into three groups of 30 participants each based on the type of sweetener used, along with a control group that will receive sucrose.

The solution will be prepared by dissolving 10 grams of the sweetener in 90 mL of distilled water and will be freshly prepared daily. A saliva sample will be collected from each participant before using the rinse, and salivary pH will be measured using a salivary pH meter. Additionally, the Streptococcus mutans count will be determined through incubation and culture.

Participants will use the mouth rinse for one minute, after which saliva samples will be collected at baseline (before rinsing), then at 1 minute, 15 minutes, and 30 minutes post-rinse. The salivary pH will be measured and recorded at each time point. The S. mutans count will be assessed before rinsing and again 30 minutes after using the solution.

ELIGIBILITY:
Inclusion Criteria:

participants aged (20-24) years.

* No active carious lesions or oral diseases.
* Generally healthy individuals without systemic illnesses.
* No prior use of preventive dental treatments

Exclusion Criteria:

* Participants currently undergoing dental treatment.
* Those taking medications that alter saliva flow.
* Presence of painful oral conditions or systemic diseases. Participants have active caries

Ages: 20 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
salivary ph measurement | Baeline salivary ph measurement (before )using mouth rinse , after 1minute , after 15 minutes , and after 30 minutes of mouth rinse
  the salivary ph will measure quantitatively using a ph meter
Streptococcus mutans count measurement | Baseline saliva collection for Streptococcus mutans count and 30 minutes after using mouth rinse saliva collection for Streptococcus mutans count
  streptococcus mutans count before mouth rinsing ,and after 30 minutes to evaluate the count if it increase or decrease

CONTACTS AND LOCATIONS:
Locations (1):
- Almustansiriyah university, Baghdad, Iraq, Iraq

IPD SHARING:
Plan to Share IPD: Undecided